CLINICAL TRIAL: NCT05903001
Title: Diaphragmatic Function as a Biomarker in Patients With Respiratory Diseases
Brief Title: Diaphragmatic Function as a Biomarker
Acronym: DFUNBIO
Status: Recruiting | Type: Observational
Sponsor: RWTH Aachen University (Other)
Responsible Party: Principal Investigator, Jens Spießhöfer, PD Dr. med., RWTH Aachen University
Other Study IDs: RWTHAachenU
Record Dates: First submitted 2023-05-18; First posted 2023-06-15 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Dyspnea; Asthmatic; COPD; Fibrosis; Pulmonary Hypertension; Asthma; Dyspnea
Keywords: dyspnea; COPD; asthma; fibrosis; pulmonary hypertension; pneumology
MeSH Terms: conditions — Dyspnea; Asthma; Pulmonary Disease, Chronic Obstructive; Fibrosis; Hypertension, Pulmonary | interventions — Electromyography; Respiration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Patients with Asthma
  Interventions: Diagnostic Test: Diaphragm Ultrasound; Diagnostic Test: Intercostal Muscle Ultrasound; Diagnostic Test: Borg scale; Diagnostic Test: MRC Breathlessness Scale; Diagnostic Test: Respiratory Questionaire; Diagnostic Test: GINA classification of Asthma; Diagnostic Test: Measurement of respiratory mouth pressure; Diagnostic Test: SNIP; Diagnostic Test: 6-minute walking distance; Diagnostic Test: 60 seconds sit-to-stand test; Diagnostic Test: Electromyography; Diagnostic Test: Lung Function
- Patients with COPD
  Interventions: Diagnostic Test: Diaphragm Ultrasound; Diagnostic Test: Intercostal Muscle Ultrasound; Diagnostic Test: Borg scale; Diagnostic Test: MRC Breathlessness Scale; Diagnostic Test: Respiratory Questionaire; Diagnostic Test: Measurement of respiratory mouth pressure; Diagnostic Test: SNIP; Diagnostic Test: 6-minute walking distance; Diagnostic Test: 60 seconds sit-to-stand test; Diagnostic Test: Electromyography; Diagnostic Test: Lung Function; Diagnostic Test: CAT-Questionnaire
- Patients with Fibrosis
  Interventions: Diagnostic Test: Diaphragm Ultrasound; Diagnostic Test: Intercostal Muscle Ultrasound; Diagnostic Test: Borg scale; Diagnostic Test: MRC Breathlessness Scale; Diagnostic Test: Respiratory Questionaire; Diagnostic Test: Measurement of respiratory mouth pressure; Diagnostic Test: SNIP; Diagnostic Test: 6-minute walking distance; Diagnostic Test: 60 seconds sit-to-stand test; Diagnostic Test: Electromyography; Diagnostic Test: Lung Function
- Patients with Pulmonary Hypertension
  Interventions: Diagnostic Test: Diaphragm Ultrasound; Diagnostic Test: Intercostal Muscle Ultrasound; Diagnostic Test: Borg scale; Diagnostic Test: MRC Breathlessness Scale; Diagnostic Test: Respiratory Questionaire; Diagnostic Test: Measurement of respiratory mouth pressure; Diagnostic Test: SNIP; Diagnostic Test: 6-minute walking distance; Diagnostic Test: 60 seconds sit-to-stand test; Diagnostic Test: Electromyography; Diagnostic Test: Lung Function; Diagnostic Test: European Society of Cardiology (ESC)/ European Respiratory Society (ERS) risk group

INTERVENTIONS:
Diagnostic Test: Diaphragm Ultrasound — Ultrasound of the Diaphragm at the end of inspiration and expiration
Diagnostic Test: Intercostal Muscle Ultrasound — Ultrasound of the Intercostal Muscles at the end of inspiration and expiration
Diagnostic Test: Borg scale — Questionnaire for Perceived Exertion (Borg Rating of Perceived Exertion Scale)
Diagnostic Test: MRC Breathlessness Scale — The MRC Dyspnoea Scale allows the patients to indicate the extent to which their breathlessness affects their mobility.
Diagnostic Test: Respiratory Questionaire — Specialized respiratory questionnaire with different domains (Emotional Domain, Dyspnea Domain, Mastery Domain, Fatigue Domain)
Diagnostic Test: GINA classification of Asthma — Patients are classified according to the GINA classification of Asthma.
  Groups: Patients with Asthma
Diagnostic Test: Measurement of respiratory mouth pressure — Inspiratory and expiratory Measurement of respiratory mouth pressure
Diagnostic Test: SNIP — Measurement of Sniff Nasal Inspiratory Pressure
Diagnostic Test: 6-minute walking distance — The maximum walking distance achieved in 6 minutes
Diagnostic Test: 60 seconds sit-to-stand test — number of repetitions achieved in sitting down and standing up in 60 seconds
Diagnostic Test: Electromyography — electromyography of the muscles of respiration via superficial electrodes
Diagnostic Test: Lung Function — Measurement of lung function via body plethysmography
Diagnostic Test: CAT-Questionnaire — COPD Assessment Test (CAT)
  Groups: Patients with COPD
Diagnostic Test: European Society of Cardiology (ESC)/ European Respiratory Society (ERS) risk group — Patients with pulmonary hypertension are classified according to the ESC/ERS risk group.
  Groups: Patients with Pulmonary Hypertension

SUMMARY:
Dyspnea is among the most common symptoms in patients with respiratory diseases such as Asthma, chronic obstructive pulmonary disease (COPD), Fibrosis, and Pulmonary Hypertension. However, the pathophysiology and underlying mechanisms of dyspnea in patients with respiratory diseases are still poorly understood. Diaphragm dysfunction might be highly prevalent in patients with dyspnea and respiratory diseases. The association of diaphragm function and potential prognostic significance in patients with respiratory diseases has not yet been investigated.

DETAILED DESCRIPTION:
The aim of the present project is to comprehensively measure respiratory muscle function and strength in patients with respiratory diseases. The investigators attempt to recruit 800 patients across four disease groups (Asthma, COPD, Fibrosis, and Pulmonary Hypertension) and the investigators intend to measure diaphragm and accessory respiratory muscle function and strength, lung function, and exercise tolerance, as well as the participants' symptom burden during one day at baseline in the investigators' lab. Thereafter, the investigators will follow up on patients by phone 3 months, 6 months, 12 months and 18 months after the investigators have seen them in the investigators' lab. In a small subset of patients (50 overall at most) and in those in whom a recently approved drug based therapy has been initiated (i.e. Sotatercept in PH, Nintedanib in ILD, Brensocatib in Bronchiectasis, Dupilumab in COPD, Anti IL-4/IL 13 or Anti IL 5 antibodies in eosinophilic asthma) follow up will not be by phone only but also in person to repeat the above mentioned non-invasive measurements. Based on these results, not only the association between dyspnea exercise tolerance and diaphragm function in patients with respiratory diseases can be assessed, but also the prognostic significance of diaphragm dysfunction in these patients can be determined. As such, hospitalization and exacerbation requiring the intake of steroids will be assessed and followed up on by phone, and therefore the prognostic significance of diaphragm dysfunction in predicting hospitalization and the intake of steroids can be determined.

ELIGIBILITY:
Inclusion Criteria:

* patient has one of the following lung diseases: COPD, bronchial asthma, pulmonary fibrosis, pulmonary hypertension
* is 18 years or older
* is mentally and physically able to understand the study and to follow instructions
* are legally competent
* signed declaration of consent

Exclusion Criteria:

* BMI > 35
* current or treatments or diseases in the past which could influence the evaluation of the study
* Expected lack of willingness to actively participate in study-related measures
* alcohol or drug abuse
* disc herniation/prolapse
* epilepsy
* wheelchair bound
* in custody due to an official or court order
* in a dependent relationship or employment relationship with investigating physician or one of their deputy
* emergency inpatient hospital stay within 4 weeks before study-specific examinations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 800 patients, 4 groups
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Dyspnea Borg scale 1 to 10 | 6 months recruiting
  Borg scale before and after "6 minute walking distance" test. Lower scores show fewer dyspnea, higher scores indicate more dyspnea.
Dyspnea Borg scale 1 to 10 | follow up 3 months after recruitment
  Borg scale before and after "6 minute walking distance" test. Lower scores show fewer dyspnea, higher scores indicate more dyspnea.
Dyspnea Borg scale 1 to 10 | follow up 6 months after recruitment
  Borg scale before and after "6 minute walking distance" test. Lower scores show fewer dyspnea, higher scores indicate more dyspnea.
Dyspnea Borg scale 1 to 10 | follow up 12 months after recruitment
  Borg scale before and after "6 minute walking distance" test. Lower scores show fewer dyspnea, higher scores indicate more dyspnea.
Dyspnea Borg scale 1 to 10 | follow up 18 months after recruitment
  Borg scale before and after "6 minute walking distance" test. Lower scores show fewer dyspnea, higher scores indicate more dyspnea.

SECONDARY OUTCOMES:
6 minute walking distance in m | 6 months recruiting
  Measurement of achieved walking distance in 6 minutes
Sit-to stand-test (60 seconds) | 6 months recruiting
  Measurement of achieved repetitions of standing up and sitting down from an initial seated position in 60 seconds.
New York Heart Association (NYHA) classification scale 1 to 4 | 6 months recruiting, follow up up to 18 months after last recruitment
  Patients are linked to a NYHA degree. Lower scores show fewer dyspnea, higher scores indicate more dyspnea.
Modified Medical Research Council (MRC) Breathlessness Scale 1 to 5 | 6 months recruiting, follow up up to 18 months after last recruitment
  Patients are assessed and grouped according to their MRC Breathlessness Scale. Lower scores show fewer dyspnea, higher scores indicate more dyspnea.
Chronic Respiratory Questionnaire (CRQ) | 6 months recruiting, follow up up to 18 months after last recruitment
  Assessments of different domains (Emotional Domain, Dyspnea Domain, Mastery Domain, Fatigue Domain) in a standardized questionnaire on a scale from 1 to 7. The scores for each question of each dimension are added together and divided by the number of completed questions in each domain. In general, higher scores mean a worse outcome and lower scores mean a better outcome.
  For the dyspnea domain for example, a high score means that patients have less dyspnea, and a low score means that patients have more dyspnea.
COPD Assessment Test (CAT-Questionnaire) from 0 to 40 points. | 6 months recruiting, follow up up to 18 months after last recruitment
  Patients are evaluated and placed into the corresponding groups. Lower scores show fewer dyspnea, higher scores indicate more dyspnea.
Global Initiative for Asthma (GINA) classification | 6 months recruiting, follow up up to 18 months after last recruitment
  Patients are assessed and grouped as mild, moderate, or severe according to the GINA classification.
Body Plethysmography | 6 months recruiting
  TLC (Total lung capacity) in percent predicted.
Diaphragm Thickening Ratio (DTR) in percent | 6 months recruiting
  Via ultrasound, the diaphragm thickening ratio (DTR) was calculated as thickness at total lung capacity (TLC) divided by thickness at functional residual capacity (FRC).
Diaphragm thickness at Total lung capacity (TLC) | 6 months recruiting
  Via ultrasound, the diaphragm thickness at TLC is measured at the maximum point of inspiration.
Diaphragm thickness at functional capacity (FRC) | 6 months recruiting
  Via ultrasound, the diaphragm thickness at FRC is measured after a normal expiration.
Diaphragm ultrasound sniff velocity in cm/s | 6 months recruiting
  Via ultrasound, the diaphragm sniff velocity was assessed during tidal breathing and following a maximum sniff.
Intercostal Muscle ultrasound thickness at Total lung capacity (TLC) in cm | 6 months recruiting
  Via ultrasound, the intercostal thickness at TLC is measured at the maximum point of inspiration.
Intercostal Muscle ultrasound thickness at functional capacity (FRC) in cm | 6 months recruiting
  Via ultrasound, the intercostal thickness at FRC is measured after a normal expiration.
Intercostal Muscle Thickening Ratio in percent | 6 months recruiting
  Via ultrasound, the intercostal muscle thickening ratio was calculated as thickness at total lung capacity (TLC) divided by thickness at functional residual capacity (FRC).
Maximum Inspiratory Pressure (MIP) in percent predicted | 6 months recruiting
  Measurement of Maximum Inspiratory Pressure
Maximum Expiratory Pressure (MEP) in percent predicted | 6 months recruiting
  Measurement of Maximum Expiratory Pressure
Sniff Nasal Inspiratory Pressure (SNIP) in percent predicted | 6 months recruiting
  Measurement of Sniff Nasal Inspiratory Pressure
Blood Gas Analysis in cmH2O | 6 months recruiting
  oxygen partial pressure (pO2)
Blood Gas Analysis in cmH2O | 6 months recruiting
  carbon dioxide partial pressure (pCO2)
Blood Gas Analysis | 6 months recruiting
  pH scale
Blood Gas Analysis in mmol/l | 6 months recruiting
  Base Excess
Blood Gas Analysis in (I1/s) percent | 6 months recruiting
  Base Excess
Electromyography (EMG) | 6 months recruiting
  Measurement of electrical activity during different breathing maneuvers (Sniff, Cough, Valsalva, Mueller) via superficial electrodes placed on the diaphragm and accessory respiratory muscles (Sternocleidomastoideus muscle, intercostal muscles).

CONTACTS AND LOCATIONS:
Overall Officials: Michael Dreher, MD, Study Director — Uniklinik RWTH Aachen; Binaya Regmi, MD, Study Chair — Uniklinik RWTH Aachen; Jens Spiesshoefer, MD, Principal Investigator — Uniklinik RWTH Aachen; Mustafa Elfeturi, Study Chair — Uniklinik RWTH Aachen; Benedikt Jörn, Study Chair — Uniklinik RWTH Aachen; Faniry Ratsimba, Study Chair — Uniklinik RWTH Aachen; Felix Wagner, Study Chair — Uniklinik RWTH Aachen; Maria Aetou, Dr. med., Study Chair — RWTH Aachen University Hospital
Locations (1):
- RWTH Aachen University Hospital, Aachen, North Rhine-Westphalia, Germany

REFERENCES:
- [Background] Daher A, Balfanz P, Aetou M, Hartmann B, Muller-Wieland D, Muller T, Marx N, Dreher M, Cornelissen CG. Clinical course of COVID-19 patients needing supplemental oxygen outside the intensive care unit. Sci Rep. 2021 Jan 26;11(1):2256. doi: 10.1038/s41598-021-81444-9. PMID 33500431
- [Background] Daher A, Balfanz P, Cornelissen C, Muller A, Bergs I, Marx N, Muller-Wieland D, Hartmann B, Dreher M, Muller T. Follow up of patients with severe coronavirus disease 2019 (COVID-19): Pulmonary and extrapulmonary disease sequelae. Respir Med. 2020 Nov-Dec;174:106197. doi: 10.1016/j.rmed.2020.106197. Epub 2020 Oct 20. PMID 33120193
- [Background] Balfanz P, Hartmann B, Muller-Wieland D, Kleines M, Hackl D, Kossack N, Kersten A, Cornelissen C, Muller T, Daher A, Stohr R, Bickenbach J, Marx G, Marx N, Dreher M. Early risk markers for severe clinical course and fatal outcome in German patients with COVID-19. PLoS One. 2021 Jan 29;16(1):e0246182. doi: 10.1371/journal.pone.0246182. eCollection 2021. PMID 33513168
- [Background] Spiesshoefer J, Henke C, Herkenrath S, Brix T, Randerath W, Young P, Boentert M. Transdiapragmatic pressure and contractile properties of the diaphragm following magnetic stimulation. Respir Physiol Neurobiol. 2019 Aug;266:47-53. doi: 10.1016/j.resp.2019.04.011. Epub 2019 Apr 25. PMID 31029769
- [Background] Spiesshoefer J, Henke C, Herkenrath S, Randerath W, Brix T, Young P, Boentert M. Assessment of Central Drive to the Diaphragm by Twitch Interpolation: Normal Values, Theoretical Considerations, and Future Directions. Respiration. 2019;98(4):283-293. doi: 10.1159/000500726. Epub 2019 Jul 26. PMID 31352459
- [Background] Spiesshoefer J, Herkenrath S, Henke C, Langenbruch L, Schneppe M, Randerath W, Young P, Brix T, Boentert M. Evaluation of Respiratory Muscle Strength and Diaphragm Ultrasound: Normative Values, Theoretical Considerations, and Practical Recommendations. Respiration. 2020;99(5):369-381. doi: 10.1159/000506016. Epub 2020 May 12. PMID 32396905